CLINICAL TRIAL: NCT03136172
Title: Observational Study on Monitoring of Systemic or Organ Blood Circulation and Perfusion for Preterm Infants
Brief Title: Monitoring of Systemic or Organ Perfusion for Preterm Infants
Status: Completed | Type: Observational
Sponsor: Inha University Hospital (Other)
Responsible Party: Principal Investigator, Juyoung Lee, Division of Neonatology, Department of Pediatrics, Inha University Hospital
Other Study IDs: Neoperfusion-2017
Record Dates: First submitted 2017-04-27; First posted 2017-05-02 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Infant, Premature; Hypoperfusion in Newborn; Necrotizing Enterocolitis of Newborn; Sepsis Newborn; Oliguria; Hypotension
MeSH Terms: conditions — Premature Birth; Neonatal Sepsis; Oliguria; Hypotension | interventions — Spectroscopy, Near-Infrared; Oximetry; Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Premature infant: premature infants with 32 weeks or less gestational age or 1,500 g or less birth weight, who born in the Inha university hospital and admit to the neonatal intensive care unit of the Inha university hospital
  Interventions: Device: NIRS (near Infra-red spectroscopy)

INTERVENTIONS:
Device: NIRS (near Infra-red spectroscopy) — 1. NIRS, INVOS 5100 cerebral/somatic oximeter monitor (Somanetics Corp, Troy, Michigan, USA)
  2. Radical-7 pulse oximeter (Masimo Corp, Irvine, CA, USA)
  3. Echocardiography (Phillips HD 15 Ultrasound system, CA, USA)
  Other Names: Pulse oximetry; Echocardiography

SUMMARY:
To investigate biomarker reflects systemic or specific organ perfusion well, we are going to the observational comparison study using several hemodynamic monitoring methods in the premature infants. It includes near-infrared spectroscopy (NIRS), pulse oximetry with perfusion index (PI) and pleth variability index (PVI) and functional echocardiography.

DETAILED DESCRIPTION:
Hemodynamic observational comparisons will be performed in 6 episodes below on each patient.

1. first 24 hours after birth
2. during red blood cell (RBC) transfusion: from 4 hours before to 4 hours after the transfusion
3. suspicion of necrotizing enterocolitis: from the suspicion point for 48 hours
4. suspicion of sepsis: from the suspicion point for 48 hours
5. oligouria (< 1 mL/kg/hour of urine): for 48 hours
6. hypotension (mean blood pressure < 30 mmHg): for 48 hours

ELIGIBILITY:
Inclusion Criteria:

* premature infants with 32 weeks or less of gestational age or 1,500 g or less of birth weight

Exclusion Criteria:

* infants without the consent of their guardians

Max Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: premature infants with 32 weeks or less of gestational age or 1,500 g or less of birth weight
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Positive predictive value of each index on hypotension | first 24 hours after birth
  Positive predictive value of each index which are recorded through the monitoring machines

CONTACTS AND LOCATIONS:
Locations (1):
- Inha University Hospital, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: No